CLINICAL TRIAL: NCT06282224
Title: Application of Augmented Reality Neuronavigation in Transnasal Endoscopic Skull Base Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: XMFHIIT-2023SL066
Record Dates: First submitted 2024-01-16; First posted 2024-02-28 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Pituitary Neoplasms
Keywords: augmented reality; Transnasal endoscopic surgery; applied research; basicranial tumor
MeSH Terms: conditions — Pituitary Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- surgery with AR-integrated endoscope (Experimental): Performing endoscopic transnasal skull base surgery with AR-integrated endoscope
  Interventions: Device: Performing endoscopic transnasal skull base surgery with AR-integrated endoscope

INTERVENTIONS:
Device: Performing endoscopic transnasal skull base surgery with AR-integrated endoscope — To explore how to use augmented reality technology (AR) to highlight important anatomical structures in the neuroendoscopic field of view, optimize the endoscopic surgical field of view, make up for the shortage of simple endoscopic field of view, make it easier for surgeons to distinguish deep anatomical structures, and reduce the intraoperative and postoperative complications of transnasal endoscopic surgery.

SUMMARY:
"For lesions in the skull base, including meningiomas, chordomas and pituitary tumors, endoscopic surgery has replaced traditional microscopes as the mainstream procedure. Although neurosurgeons can enlarge the surgical area using a neuroendoscope, it does not provide any information on the morphology and location of anatomical structures beneath visible surfaces. Due to the complex anatomical relationships of adjacent structures in the skull base, lesions occurring here are often located deep within anatomy that is difficult to fully expose and remove with endoscopic surgery alone. Especially when dealing with larger tumors that surround major arteries and nerves, limited visibility at surface level can easily damage blood vessels or nerves causing complications such as bleeding during or after surgery, deformities or functional impairments. The purpose of this study is to explore how augmented reality (AR) technology can highlight important anatomical structures in a neuroendoscope's field of view to optimize surgical visibility beyond what is possible with just an endoscope alone. This will make it easier for surgeons to distinguish deeper anatomical structures and reduce intraoperative and postoperative complications associated with endoscopic surgery."

DETAILED DESCRIPTION:
1. Research protocol The surgical AR neuroendoscopic system in this study mainly includes three core links: (1) virtual image or environmental modeling. AR systems use data derived from color or texture differences between anatomical structures in CT or MRI tomography, as well as whole-brain angiography, to complete a 3D reconstruction of a subsurface target in a computer. This process can also be done manually using the 3D-Slicer software. (2) Registration of virtual environment and real space. Registration technology is essential for AR systems, as it enables real-time tracking of anatomical structures in the endoscopic field of view. Registration can be done by a variety of means, such as the 3D Cartesian system, which is based on framing technology, which can determine the position and attitude of the imaging device, while also allowing the virtual environment to make rapid changes and register when the position changes in the real world. Or use frameless registration to register virtual match points with known anatomical landmarks in real space. (3) The final demand is to combine the virtual environment with the real environment to display technology. It can be divided into head-mounted display (HMD), enhanced external display, enhanced optical system, enhanced window display and image projection. Using HMDs to overlay virtual environments with video feeds from real environments (video perspective). Utilize a simple, stand-alone screen as an enhanced display to display virtual content on a video originating from a neuroendoscope.

After the above links are successfully achieved, transnasal skull base surgery is performed using neuroendoscope with AR to achieve real-time tracking, accurately identify anatomical structures, and reduce the risk of neurovascular injury and complications in skull base surgery.

Subjects: About 100 cases of neuroendoscopic skull base surgery performed in the Department of Neurosurgery of the First Affiliated Hospital of Xiamen University, regardless of gender and age.

Inclusion Criteria: 1. Patients undergoing transnasal endoscopic skull base surgery in our department. 2. Thin-slice head MRI and CTA scans were performed before surgery. Exclusion Criteria: 1. Patients without clear preoperative imaging data. 2. Patients who do not agree to receive AR fusion neuroendoscopic assistance. 3. Patients with incomplete medical records.

Intervention: Participants were divided into two groups to undergo transnasal skull base surgery using common neuroendoscopy and neuroendoscopy infused with augmented reality technology and compared.

Evaluation methods: The surgical effect was evaluated according to the patient's tumor size, pathological type, operation time, length of hospital stay, complications, and whether there was a history of pituitary surgery.

Effectiveness evaluation indicators (primary efficacy index and secondary efficacy index):

The main efficacy indicators: duration of surgery, whether the augmented reality navigation was successfully established during the operation, whether the augmented reality navigation was accurate during the operation, the incidence of cerebrospinal fluid leakage during the operation, and the incidence of damage to important anatomical structures during the operation Secondary efficacy measures: endocrine improvement rate, visual field improvement rate, length of hospital stay, etc.

Statistical methods: Chi-square test was used for counting data, t-test was used for measurement data, and SPSS software was used for data processing.

Participant participation time: one year after the patient is admitted to the hospital to be discharged.

Location: The First Affiliated Hospital of Xiamen University Hypothesis: Neuroendoscopy integrated with augmented reality technology can greatly promote intraoperative orientation and facilitate the surgeon's observation of correlation anatomy. Therefore, we hypothesize that neuroendoscopy with augmented reality technology can reduce surgical complications and improve surgical efficacy compared with traditional endoscopy.

All eligible subjects were randomly divided into two groups to undergo traditional nasal endoscopic surgery and endoscopic transnasal surgery with augmented reality technology, and relevant data were collected for statistical analysis after the surgery. None of the subjects were grouped before surgery. Traditional transnasal endoscopic surgery was used as the control group to evaluate the therapeutic effect of augmented reality endoscopy. Before the study was carried out, the research group had a comprehensive grasp of the factors such as the size of the cases requiring nasal surgery and the age and gender composition of the patients who needed to undergo nasal surgery in our hospital, established a good sampling framework, and strictly implemented stratified and proportional sampling, so as to avoid and reduce selective bias. The research team has done a good job of coordination and mobilization before the investigation, obtained the cooperation of the department and the relevant departments of the outpatient department, established a trust relationship with the patients, reduced the refusal of visits, thereby reducing the selectivity bias, and can improve the authenticity of the interviews and reduce the bias of information. Avoid and reduce refusals as much as possible. This study followed ethical principles throughout the process, obtained the trust and cooperation of patients, and avoided and reduced information bias. Responsible and communicative team members were selected as investigators to reduce information bias.

The duration of this study was from the time the patient was admitted to the hospital and the patient was discharged 1 month later, with an average of about 1 month. The follow-up time was 1 month, 3 months, 6 months and 1 year after surgery, respectively.

The main intervention method in this study was to use a neuroendoscope developed by the research group integrating augmented reality technology instead of traditional neuroendoscopy for transnasal skull base surgery.

Study endpoint: The study endpoint is reached if the study subject completes all phases of the study and follow-up according to the study protocol or withdraws the informed consent.

Sample size: A total of 100 cases of AR fusion neuroendoscopic transnasal skull base lesion surgery were completed in 3 years. The expected loss-to-follow/drop-out rate is less than 5%.

Study intervention: Transnasal skull base surgery using an augmented reality neuroendoscope developed by the research group instead of a traditional endoscope, which utilizes the hospital's existing Medtronic S7 navigation and Carl STORZ endoscope, and the safety of the above devices has been validated. The surgical instruments used to complete all cases are the same model of the same brand and the same operator, so as to avoid affecting the surgical process due to hardware reasons and manual operation. For each completed operation, the patient's relevant imaging information will be backed up, and the patient's case number will be recorded to prevent the loss of case information. The registration of intraoperative endoscope and AR was in accordance with the operating procedures, and after the registration was completed, the body surface markers were used to ensure the authenticity and accuracy of intraoperative AR images. At the time of discharge, all cases were informed of regular outpatient re-examination and postoperative follow-up. The case data is summarized once a month, and a special person is responsible for keeping the summary. The research team is cooperating and has rich experience in surgery. We have a professional operating room team to ensure the smooth progress of the operation. AR navigation may cause errors during the registration process, which should be operated in strict accordance with the navigation operation procedure, and in vitro navigation tests using body surface landmarks to reduce errors before performing surgery, and iCT registration should be used if necessary. In all cases, 4 CT scans of the head, 2 CT scans of the chest, 3 sMRI scans of the brain, 4 blood draws, and 1 bedside electrocardiogram were planned. If necessary, routine preoperative examinations such as color ultrasound and Holter electrocardiogram are performed. All surgical instruments are sterilized and packaged by the Supply Room of the First Affiliated Hospital of Xiamen University. All surgical equipment All of them are stored in a cool and dry place in the operating room of the First Affiliated Hospital of Xiamen University, and are adjusted and regularly maintained by professional engineers. The use of neuroendoscopy, neuronavigation and other devices is in accordance with the instructions and guidelines.

Measures to reduce bias: data and data collection should be as precise and precise as possible, and appropriate statistical methods should be selected.

Follow-up and compliance: A total of 4 follow-up visits were performed at 1 month, 3 months, 6 months and 1 year after surgery. During the follow-up, CT/MRI of the head was taken, blood tests were taken, and endocrine functions such as thyroid and pituitary gland were checked. By establishing a relationship of trust with patients in advance, improving service attitude, optimizing the treatment process, strengthening preoperative and postoperative guidance, and reminding patients to review in a timely manner, patients can improve their compliance.

Study Intervention Commitment:

Using the existing Medtronic S7 navigation and Carl STORZ endoscope to develop AR technology, the use of all equipment follows the instructions and guidelines, and the whole process of the operation is videotaped, and the postoperative review is carried out by a special person to ensure the smooth implementation of the surgical process, all the doctor's orders and medications during the patient's stay in the hospital are supervised by a special person, and the influence of medical drugs and operations on the surgical results is excluded. Medical records and other medical documents are kept by the research team, and the patient review reminder and follow-up are carried out by the special person.

Suspension of study intervention: If a large number of the following serious adverse reactions occur during the course of the study, the trial will be discontinued after the comprehensive decision of the investigator. (1) Severe cerebrospinal fluid rhinorrhea complications (2) Symptoms of periorbital bruising and hematoma in the eye, or severe vision loss, blurred vision and other manifestations. (3) Severe nasal bleeding, causing anemia or even shock, or nasal adhesions, which seriously affects nasal ventilation and sinus drainage. (4) Damage to large blood vessels and nerves, (5) Severe symptoms of endocrine disorders, (6) Severe cerebral edema or intracranial infection During the study interruption: carefully check the software and hardware problems of the endoscopy system, check the accuracy of the image output, and test the effectiveness of the software. Check whether there are any problems with the surgical conditions, surgical instruments and surgical team. and provide effective medical assistance to subjects who have adverse events. The relevant information of all subjects with adverse events was collected, including but not limited to: age, gender, time of consultation, image number, diagnosis, visual field, endocrine status, operation time, whether there was cavernous sinus hemorrhage during the operation, whether the tumor was completely resected, whether there was cerebrospinal fluid leakage, whether the augmented reality navigation was successfully established during the operation, whether the augmented reality navigation was accurate during the operation, the length of hospital stay, the postoperative visual field, and the endocrine situation.

Withdraw/Withdraw from the Study Subject: The investigator may suspend or withdraw the study subject if the study subject has: (1) pregnancy (2) significant non-compliance with the study intervention (3) if there are clinical side effects, abnormal laboratory tests, or other clinical conditions that make continued participation in the study no longer in the best interest of the study subject (4) disease progression that necessitates discontinuation of the study intervention (5) the study subject meets the exclusion criteria (new or confirmed) (6) the study subject cannot receive the study intervention for a certain period of time (7) the study subject who signs the informed consent form, is randomized, but does not receive the study intervention will be replaced. Study subjects who have signed informed consent, randomized, received study intervention, and subsequently withdrawn will be or will not be replaced.

Loss to follow-up: The follow-up period for this study is 1 year from the date of discharge of the patient, and can be considered lost to follow-up when the study subject stops the scheduled study follow-up, cannot complete the study-specified procedures, or the investigator cannot contact the study subject. The loss rate was reduced by recording a variety of contact information such as telephone number and email address during subject registration, arranging a special person in the research group to be responsible for reminding subjects to review and follow-up regularly, designing a stable population to facilitate follow-up, increasing sample size, and reducing the impact of loss to follow-up.

Observation items and testing time points: During the subject screening period, ensure that each subject has an indication for surgery, and there are no contraindications to surgery. Random sampling, stratified sampling, and confidentiality of the results were kept to the subjects when grouping. During the intervention period, various examination indicators and imaging data were collected for the subjects before surgery, 3D modeling was used for preoperative planning, the accuracy of the 3D model was verified during the operation, and the surgical operation was performed with augmented reality endoscopy, and the examination results were collected after surgery to evaluate the surgical effect. During the follow-up period, telephone follow-up or face-to-face consultations were conducted at one month, three months, six months and one year after surgery to further evaluate the efficacy of surgery. Finally, the medical record data were summarized, and the efficacy of the augmented reality neuroendoscope developed by the research group was evaluated after statistical analysis.

Efficacy Evaluation Criteria:

1. Evaluation of surgical efficacy:

   Effectiveness evaluation indicators: including but not limited to age, gender, time of consultation, image number, diagnosis, operation time, whether the tumor is completely resected, whether the augmented reality navigation is successfully established during the operation, whether the augmented reality navigation is accurate during the operation, and the length of hospitalization.

   Safety evaluation: preoperative visual field, endocrine condition, intraoperative cavernous sinus hemorrhage, cerebrospinal fluid leakage, postoperative visual field, endocrine condition, etc.
2. Comprehensive efficacy evaluation: postoperative patient satisfaction, operator satisfaction, etc.

Observation of adverse events: Adverse events refer to a series of malignant events that may occur in patients during neuroendoscopic surgery, including but not limited to endoscopic burns, endoscopic mechanical injury, contamination caused by endoscope detachment, intraoperative neurovascular injury, intraoperative awakening and awareness, postoperative cerebrospinal fluid leakage, postoperative nursing negligence, etc.

Monitoring of adverse events: mainly through manual monitoring, manual and electronic composite monitoring, and automatic monitoring system. The recording, handling and reporting of adverse events should follow the following principles: 1. Establish an adverse event reporting system. 2. Respond in time to reduce losses. 3. Treat fairly, focusing on the system rather than the individual. 4. Establish a mechanism for discussing errors. 5. Analyze feedback, share information, and enhance collaboration among researchers 6. Follow up and implement, strengthen management, and strengthen quality control of the research process 7. Continuous improvement, prevent recurrence, and continuously optimize the research process.

Quality control and quality assurance of the study: 1. The surgical instruments used to complete the operation in all cases are the same model of the same brand, and the surgeon is the same person, so as to avoid affecting the surgical process due to hardware reasons and human operation. 2. For each completed operation, the patient's relevant imaging information will be backed up, and the patient's case number will be recorded to prevent the loss of case information. 3. The registration of the intraoperative endoscope and AR is in accordance with the operating procedures, and the body surface markers are used for examination after the registration is completed to ensure that the intraoperative AR images are true and accurate. 4. Inform all cases of regular outpatient review at the time of discharge, and maintain postoperative follow-up. 5. Summarize the case data once a month, and a special person is responsible for keeping the summary. 6. The department has a large number of surgeries, and there are a variety of cases for study.

Pre-assessment of project risk and risk disposal plan: All surgeries will be performed by professionals such as surgeons, with tacit cooperation with the research team, rich surgical experience, and a professional operating room team to ensure the smooth progress of the operation. Theoretically does not increase any risk to the subject. However, in the course of routine clinical diagnosis and treatment, once there is any discomfort, the professional doctors in the research group will give reasonable further treatment to the subjects.

The surgical instruments used to complete all cases are the same model of the same brand, and the surgeons are all the same person, so as to avoid affecting the surgical process due to hardware reasons and human operation.

For each completed operation, the patient-related imaging information will be backed up, and the patient's case number will be recorded to prevent the loss of case information.

The registration of intraoperative endoscope and AR was in accordance with the operating procedures, and after the registration was completed, the body surface markers were used to ensure the authenticity and accuracy of intraoperative AR images.

At the time of discharge, all cases were informed of regular outpatient re-examination and postoperative follow-up. The case data is summarized once a month, and a special person is responsible for keeping the summary.

Data security monitoring: Clinical research will develop a data security monitoring plan based on the size of the risk. All adverse events are recorded in detail, properly handled and tracked until properly resolved or the condition is stable, and the ethics committee, competent department, Sponsors and drug regulatory authorities report serious adverse events and unexpected events, etc., the principal investigator regularly conducts cumulative reviews of all adverse events, and holds investigator meetings to evaluate the risks and benefits of the study if necessary, double-blind trials can be urgently unblinded if necessary to ensure the safety and rights of subjects, independent data monitors will be arranged to monitor the study data for studies with greater than minimum risk, and independent data security supervision will be established for high-risk studies The committee monitors the accumulated safety data as well as the efficacy data to make recommendations on whether or not to proceed with the study.

XIII. Statistical Processing Statistical analysis was performed using SPSS 22.0 software (SPSS Inc., Chicago, IL). Quantitative data were described as mean and range. Qualitative data are described by numbers, rates, and ratios. The normality of the data was tested using the Kolmogorov-Smirnov test. For continuous variables, if the data are normally distributed, the t-test was used for comparison between the two groups. If the data distribution is asymmetrical, the Mann-Whitney U test is used. The chi-square test was used for the analysis of discontinuous variables. The diagnostic performance of the CAC test was assessed by constructing receiver operating characteristic (ROC) curves and calculating the area under the curve (AUC). All statistical tests were bilateral, and significance was set to P < 0.05 and 95% CI.

2. Research Objectives Main objectives: To explore the solution of integrating AR technology in the interface of neuroendoscopic view, and use this technology to complete transnasal and skull base surgery, which is difficult to perform endoscopic surgery alone Secondary objectives: To provide a reference for the development of new functions of neuroendoscopy.

ELIGIBILITY:
Inclusion Criteria：

* Patients who are suitable for Transnasal endoscopic surgery 。
* Patients who have performed thin-layer head MRI and CTA scans before surgery.

Exclusion Criteria：

* Patients without clear preoperative imaging data.
* Patients who do not agree to receive the assistance of AR fusion neuroendoscopy.
* Patients with incomplete medical records.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2025-01-11 (Estimated); Study Completion 2026-01-11 (Estimated)

PRIMARY OUTCOMES:
Postoperative Recovery of Transnasal Surgery | at the time points of baseline，3 months, 6 months and 1 year after surgery
  Observe whether the preoperative symptoms (including endocrine abnormalities, impaired visual field, headache, etc.) were alleviated after surgery.
Postoperative complication | at the time points of baseline，3 months, 6 months and 1 year after surgery
  Postoperative complication including cerebrospinal fluid leakage, significant neurovascular injury, visual impairment, endocrine disorders, nasal septum perforation and postoperative diabetes insipidus.

CONTACTS AND LOCATIONS:
Overall Officials: Hongwei Zhu, doctorate, Study Director — The First Affiliated Hospital of Xiamen University
Locations (1):
- The First Affiliated Hospital of Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: Obtain data immediately after publication，indefinite duration
Access Criteria: anyone